CLINICAL TRIAL: NCT00348582
Title: Acular LS vs. Nevanac in Post op Inflammation Following Cataract Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 5217
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2007-06-25 (Estimated); Status verified 2007-06

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Ketorolac; nepafenac

INTERVENTIONS:
Drug: Ketorolac, Nepafenac

SUMMARY:
The purpose of this study is to compare the clinical outcomes, safety and efficacy in patients randomized to receive either ketorolac or nepafanac following cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* · Male or female > 18 years of age scheduled to undergo cataract surgery

  * Must be in good general health. Patients with systemic diseases will be enrolled only if there are no ocular manifestations of their disease (ie diabetics with normal retinal exams)
  * Ability to provide informed consent and likely to complete all study visits

Exclusion Criteria:

* · Known contraindication to any study medication or any of their components

  * Uncontrolled systemic disease
  * Required use of ocular medications other than the study medications during the study
  * Abnormal pre-operative OCTs if obtainable
  * Diabetic patients
  * Use of oral NSAIDS
  * Patients with ocular disease (macula degeneration, glaucoma, corneal disease) which reduces the potential visual rehabilitation (patients will ocular disease that will no preclude achievement of a 20/20 visual outcome may be included)..

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Francis Mah, MD, Principal Investigator — University Pittsburgh Medical Center Eye and Ear Institute
Locations (1):
- Dr. Francis, Pittsburgh, Pennsylvania, United States